CLINICAL TRIAL: NCT00641355
Title: Acute Phase Proteins as Early Markers in Sepsis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Zurich (Other)
Responsible Party: PD Dr. Marius Keel, University Hospital of Zurich
Other Study IDs: StV 26-2007
Record Dates: First submitted 2008-03-17; First posted 2008-03-24 (Estimated); Last update posted 2008-03-24 (Estimated); Status verified 2008-03

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: No intervention — No intervention

SUMMARY:
Monitoring of different serumproteins after severe trauma and during trauma-induced sepsis.

* Trial with surgical intervention

ELIGIBILITY:
Inclusion criteria:

* Patients with severe trauma (ISS score > 16), both genders, patients on ICU

Exclusion criteria:

* Moribund patients (pH <7,1, lactate >15mmol, Basedeficit > 15mEq/L, severe heart or liver injuries, GCS never over 5 after trauma)
* Severe head injuries (AIS head >4)
* Patient with severe infectious diseases, or diseases which severely affect the immune system (diabetes, Alkohol or nicotine abuse)
* Non-german speaking patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe trauma
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2008-04; Study Completion 2012-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland